CLINICAL TRIAL: NCT04574960
Title: Neoadjuvant Chemotherapy in Upper Tract Urothelial Cancer: A Multicentre, Feasibility Pilot Trial
Brief Title: Neoadjuvant Upper Tract Invasive Cancer Trial (NAUTICAL)
Acronym: NAUTICAL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Bladder Cancer Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-5149
Record Dates: First submitted 2020-09-18; First posted 2020-10-05 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer; Bladder Urothelial Carcinoma
Keywords: Upper tract urothelial carcinoma; UTUC
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant Chemotherapy Arm (Experimental): Gemcitabine/Cisplatin will be administered on a 3-week cycle for up to 4 cycles. This will be followed by surgical intervention (nephroureterectomy or ureterectomy).
  Interventions: Drug: Gemcitabine; Drug: Cisplatin
- Adjuvant Chemotherapy Arm (Standard of Care) (Active Comparator): Patients will undergo surgical intervention (nephroureterectomy or ureterectomy) followed by adjuvant chemotherapy.
  Patients with a GFR greater or equal to 60 mL/min will receive Gemcitabine/Cisplatin while those with a GFR greater or equal to 30 mL/min but less than 60 mL/min will receive Gemcitabine/Carboplatin.
  Gemcitabine/Cisplatin will be administered on a 3-week cycle for up to 4 cycles.
  Gemcitabine/Carboplatin will be administered on a 3-week cycle for up to 4 cycles.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2, IV infusion on days 1 and 8 of each 3-week cycle
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin 70 mg/m^2, IV infusion on day 1 of each 3-week cycle
  Other Names: Platinol
Drug: Carboplatin — Carboplatin AUC 5-6 calculated using the Calvert formula on day 1 of each cycle
  Other Names: Paraplatin
  Arms: Adjuvant Chemotherapy Arm (Standard of Care)

SUMMARY:
Upper tract urothelial cancer (UTUC) is cancer in the lining of the kidney or ureter (the tube that drains the kidney). This type of cancer is rare and as a result, there are only a few studies that have looked at it.

Standard of care for UTUC would be surgery followed by chemotherapy (adjuvant chemotherapy). However, we know from studies that have looked at cancer of the lining of the bladder, which is a similar cancer in many ways, that treating people with chemotherapy before surgery (neoadjuvant chemotherapy) can lead to longer survival compared to the standard of care. There are no studies to show this in UTUC. Neoadjuvant chemotherapy is thought to help improve survival by treating any cancer that may have spread from the original tumour but that is not visible yet on scans. This study would be the first clinical trial in Canada to evaluate the use of chemotherapy before surgery in this disease setting.

Since UTUC is rare, the purpose of this study is to determine if it is possible to enrol enough patients to a trial looking at the use of chemotherapy before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed radiographically visible (CT or MRI) cT1-4 N0 M0 with positive selective urinary cytology, positive bladder urinary cytology, or endoscopic biopsy for high grade urothelial cell carcinoma
* Age ≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) score 0-1
* Medically appropriate candidate for radical nephroureterectomy or ureterectomy as per participating site attending urologic oncologist
* Medically appropriate candidate for cisplatin-based chemotherapy as per participating site attending medical oncologist
* Adequate organ system function defined as follows: absolute neutrophil count ≥ 1500/mm3, platelets ≥ 100,00/mm3, hemoglobin ≥ 90 g/L, ALT and AST < 2.5 x upper limit of normal, electrolytes (Na, K, Mg, Ca): within normal limits, GFR ≥ 60 mL/min

Patients who are randomized to the adjuvant chemotherapy will be reassessed for suitability to receive adjuvant chemotherapy after definitive surgery (nephroureterectomy or ureterectomy) based on the following criteria:

* pT2-4 N0-3 M0 or pT any N1-3 M0 with predominant urothelial component
* ECOG score 0-2
* Medically appropriate candidate for platin-based chemotherapy as per participating site attending medical oncologist
* Adequate organ system function defined as follows: absolute neutrophil count ≥ 1500/mm3, platelets ≥ 100,00/mm3, hemoglobin ≥ 90 g/L, ALT and AST < 2.5 x upper limit of normal, electrolytes (Na, K, Mg, Ca): within normal limits, GFR ≥ 30 mL/min

Exclusion Criteria:

* Metastatic disease
* Radiographically visible nodal disease
* Concurrent muscle-invasive bladder cancer (non-muscle invasive bladder cancer is acceptable)
* Solitary kidney
* Other cancer diagnosis or systemic chemotherapy use within 2 years of study enrollment (prior bladder cancer and intravesical therapy allowed)
* Concomitant diseases that are a formal exclusion to cisplatin chemotherapy (deafness, ≥ grade II neuropathy, serious active infection)
* Concomitant use of any other investigational drugs
* Pregnancy or breast feeding (you must remain on contraception, not father a child or donate sperm while receiving gemcitabine/cisplatin and for 6 months following the last dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrolling cT1-4N0 M0 UTUC patients in a randomized trial of neoadjuvant chemotherapy versus standard of care by assessing pilot trial recruitment rates | 24 months
Disease-free survival (DFS) | 36 months
  DFS is defined as the time from randomization to development of intravesical recurrence, contralateral upper tract recurrence or distant metastasis
Rate of complete pathologic response | 36 months
  Complete pathologic response is defined as pT0 N0

SECONDARY OUTCOMES:
Site-specific enrolment rate | 24 months
Number of patients approached per site per month | 24 months
Number of patients randomized per site per month | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Girish Kulkarni, MD, Principal Investigator — University Health Network - Princess Margaret Hospital
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario